CLINICAL TRIAL: NCT01976832
Title: Music-with-Movement Intervention for People With Early Dementia and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Claudia K Y Lai, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5-ZH96
Record Dates: First submitted 2013-10-23; First posted 2013-11-06 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Dementia; Anxiety; Sleep; Depression; Quality of Life
MeSH Terms: conditions — Dementia; Anxiety Disorders; Depression | interventions — Movement; Drug Interactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music with movement (Experimental): Participants in the intervention group will receive the intervention delivered by their family member according to the validated 8-weeks music with movement (MWM) intervention protocol.
  Interventions: Behavioral: Music with movement
- Social interaction (Active Comparator): The control group will receive a protocol for social interaction as the control condition, where caregivers were asked to discuss up to date news with PWeD.
  The design of the control condition will be highly similar to the MWM protocol in terms of the frequency and duration of the sessions, the number of people involved, and the total intervention period.
  Interventions: Behavioral: Social interaction

INTERVENTIONS:
Behavioral: Music with movement — Participants in the intervention group will receive the intervention delivered by their family member according to the validated 8-week music with movement (MWM) intervention protocol.
  Arms: Music with movement
Behavioral: Social interaction — The control group will receive a protocol for social interaction as the control condition, where caregivers were asked to discuss up to date news with PWeD.
  The design of the control condition will be highly similar to the MWM protocol in terms of the frequency and duration of the sessions, the number of people involved, and the total intervention period.
  Arms: Social interaction

SUMMARY:
This study intends to use music and movement (MWM) to reduce anxiety and behavioral symptoms of people with early dementia (PWD) and their family carers in the community. It also aims to examine whether MWM can enhance the sleep quality of PWD and their family caregivers and promote their well-being.

This is a mixed methods study with the quantitative paradigm being the main research approached used. The quantitative arm will be a randomized controlled trial (RCT). The qualitative arm will adopt a naturalistic approach through interviewing for data collection. Recruited subjects from the community centres of non-government organizations (NGOs) will be randomly allocated to the intervention and control group.

The outcome measures of the PWD will include Rating Anxiety in Dementia (RAID), Geriatric Depression Scale (GDS), Neuropsychiatric Inventory Questionnaire (NPI-Q), Pittsburgh Sleep Quality Index (PQSI), Quality of Life - Alzheimer's Disease (QOL-AD), Mini-Mental State Examination (MMSE), Revised Life Event Scale (RLES), Modified Brathel Index (MBI) and Non-pharmacological Therapy Experience Scale (NPTES), whereas the outcome measures of the family caregivers will be Patient Health Questionnaire 9 (PHQ-9), Generalized Anxiety Disorder 7 (GAD-7), Zarit Burden Scale (ZBD), Pittsburgh Sleep Quality Index (PSQI), Reverse Life event Scale (RLES), and World Health Organization Quality of Life-BREF (WHOQOL-BREF).

To address the research questions, data will be collected at baseline (T0), immediately post-intervention at 8-weeks (T1), and 8 post-intervention (T2). The qualitative arm of this study will contribute to the understanding of issues and effects of MWM as an intervention. Its finding will complement the results obtained from the RCT.

ELIGIBILITY:
Inclusion Criteria:

1. PWD

   * Aged 65 or above
   * Community-dwelling
   * With early dementia [Clinical Dementia Rating (CDR) Scale scored between 0.5 to 1, denoting mild to early signs of cognitive impairment]
   * In a stable medical condition
   * Communicate in Cantonese
   * Has a family caregiver who is willing to participate in the study
2. Family caregiver of the recruited PWD

   * Is the primary caregiver of the PWD (defined as the one in the family who is responsible for taking care of the PWD regardless of whether s/he is living together with the PWD in the same dwelling place. That is to say, him/herself considers self as the person responsible to provide needed care for the PWD; or other family members would expect him/her to perform or be responsible for main caregiving tasks needed by the PWD.)
   * Is related to the PWD and not a paid live-in care attendant
   * Paid caregiver is allow to assist the primary caregivers if he/she attended the MWM training, but can contribute no more than 50% of the delivery of intervention.
3. Staff

   * Completed no less than 80% of the training program for delivery the MWM protocol
   * Has been involved in the delivery of the MWM intervention to the intervention group for at least one cycle of recruitment Note: staff recruitment as the informant of the qualitative arm of this study is also entirely voluntary.

Exclusion Criteria:

1. PWD With acute exacerbation of chronic illnesses that affects the adherence of the MWM protocol, e.g., acute heart failure, relapse of acute depressive disorder unable to hear even with the use of hearing aids unable to sit independently for around 45 minutes
2. Family caregivers of the recruited PWD

   - Nil
3. Staff - Nil

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change of Rating anxiety in Dementia (RAID) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1

SECONDARY OUTCOMES:
Change of Geriatric Depression Scale (GDS) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Neuropsychiatric Inventory Questionnaire(NPI-Q) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Pittsburgh Sleep Quality Index (PQSI) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD and Caregivers of PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Quality of Life - Alzheimer's Disease (QOL-AD) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Patient Health Questionnaire 9 (PHQ-9) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For Caregivers of PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Zarit Burden Scale (ZBS) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For Caregivers of PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of World Health Organization Quality of Life-BREF (WHOQOL-BREF) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For Caregivers of PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Generalized Anxiety Disorder 7 | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For Caregivers of PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Mini-Mental State Examination (MMSE) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Revised Life Event Scale (RLES) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD and Caregivers of PWD
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Lawton's Instrumental Activity of Daily Living (IADL) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1
Change of Modified Barthel Index (MBI) | At baseline (T0), immediately post-intervention at 8-weeks (T1), and 8-weeks post-intervention (T2)
  For PWD only
  Comparisons of changes of RAID will be considered as follows:
  1. T1 - T0
  2. T2 - T0
  3. T2 - T1

OTHER OUTCOMES:
Change of Non-pharmacological Therapy Experience Scale (NPTES) | once per month within the intervention period
  NPTES will be collected within the intervention period on several occasions. That is to say, to be obtained once per month between T0 to T1, and only for the intervention group. It is an observational tool intended for capturing the qualitative information during an intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kam Yuk, Claudia Lai, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; Shuk Ching, Jacqueline Ho, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; Sze Ki, Daphne Cheung, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai CK, Lai DL, Ho JS, Wong KK, Cheung DS. Interdisciplinary collaboration in the use of a music-with-movement intervention to promote the wellbeing of people with dementia and their families: Development of an evidence-based intervention protocol. Nurs Health Sci. 2016 Mar;18(1):79-84. doi: 10.1111/nhs.12238. Epub 2015 Sep 10. PMID 26354593